CLINICAL TRIAL: NCT07300410
Title: Usability, Acceptance, and Effectiveness of a Coach-Guided, App-Based Mental Health Intervention: The beWell Tirol Pilot Study
Brief Title: App-Based Coaching Program to Improve Mental Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BeWell271125
Record Dates: First submitted 2025-11-27; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Psychological Distress
Keywords: Digital Mental Health; App-Based Intervention; Cognitive Behavioral Therapy (CBT); Psychological Distress; Coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- beWell Tirol Intervention (Experimental): A 4-month digital mental health program delivered via the beWell Tirol app. The intervention includes psychoeducation, cognitive-behavioral exercises, interactive tools, digital diaries, and bi-weekly video coaching.
  Interventions: Device: Digital Mental Health Program with Coaching

INTERVENTIONS:
Device: Digital Mental Health Program with Coaching — This intervention is a 4-month digital mental health program with coaching. Participants use a mobile app that provides access to psychoeducational content, interactive cognitive-behavioral exercises, digital diaries, and self-monitoring tools. The program includes individualized exercise selection, where participants choose exercises every two weeks in collaboration with a trained coach. The intervention also incorporates bi-weekly 20-30 minute video coaching sessions, delivered within the app, to support motivation, clarify questions, and tailor the training plan. Exercises include relaxation techniques, mindfulness exercises, positive psychology activities, journaling tools, daily structuring tasks, and problem-solving strategies.

SUMMARY:
The goal of this clinical trial is to learn if a coach-guided, app-based mental health program can improve well-being and reduce psychological distress in adults experiencing elevated stress levels. The main questions it aims to answer are:

* Does the beWell Tirol program show high usability and participant satisfaction?
* Does participation in the program lead to improvements in psychological distress, resilience, self-efficacy, coping strategies, emotion regulation, and quality of life?

Participants will:

* Complete a 4-month digital mental health program using the beWell Tirol app
* Attend bi-weekly video coaching sessions with a trained psychologist
* Choose individualized cognitive-behavioral exercises within the app
* Complete questionnaires at baseline, post-intervention, and 3-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Living in Tyrol (Austria) or South Tyrol (Italy)
* Elevated psychological distress (Brief Symptom Inventory / BSCL Global Severity Index T-score > 60 based on age and gender)
* Sufficient German language skills to use the app and complete questionnaires
* Access to a smartphone or tablet and the internet
* Willing and able to participate in the 4-month digital program and follow-up assessments
* Provided written informed consent

Exclusion Criteria:

* Non-German-speaking individuals
* Acute psychiatric crisis or acute suicidality requiring immediate face-to-face treatment
* Any condition that, in the judgment of the investigators, would prevent safe participation or the completion of the app-based intervention (e.g., severe cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-01-13 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Usability of the digital mental health program | Right after the intervention ended
  Usability will be assessed using the System Usability Scale (SUS), a 10-item validated questionnaire measuring perceived usability of digital systems. Scores range from 0 to 100, with higher scores indicating better usability.

SECONDARY OUTCOMES:
Participant satisfaction | Right after the intervention ended
  Satisfaction will be measured using a 10-item participant satisfaction questionnaire assessing overall satisfaction, perceived usefulness, impact on well-being, and coach satisfaction. Items are rated on a 4-point Likert scale (strongly disagree to strongly agree). Higher scores indicate greater satisfaction.
Psychological distress | Baseline, right after the intervention ended, 3-month follow-up
  Psychological distress will be measured with the Perceived Stress Scale (PSS-10), which assesses whether individuals perceive situations in their lives as excessively uncontrollable and overwhelming. Scores ranging from 0 to 13 indicate low stress, scores ranging from 14 to 26 indicate moderate stress, and scores ranging from 27 to 40 indicate high perceived stress.
Resilience | Baseline, right after the intervention ended, 3-month follow-up
  Resilience will be assessed using the RS-13 Resilience Scale, a 13-item measure with scores ranging from 13-91. Higher values reflect greater resilience.
Self-efficacy expectation | Baseline, right after the intervention ended, 3-month follow-up
  Self-efficacy will be measured using the General Self-Efficacy Scale (SWE), consisting of 10 items rated on a 4-point Likert scale. Higher scores indicate greater perceived self-efficacy.
Emotion regulation | Baseline, right after the intervention ended, 3-month follow-up
  Emotion regulation will be measured using the Emotion Regulation Questionnaire (ERQ), including the subscales Cognitive Reappraisal (6 items) and Expressive Suppression (4 items). Higher scores reflect greater use of the respective strategy.
Quality of Life: WHOQOL-BREF Global Score | Baseline, right after the intervention ended, 3-month follow-up
  Quality of life will be assessed using the WHOQOL-BREF, comprising four domains: physical health, psychological health, social relationships, and environment. Higher scores reflect better quality of life.
Coping strategies | Baseline, right after the intervention ended, 3-month follow-up
  Coping will be assessed using the SVF-ak 42, measuring positive and negative coping responses. Subscale scores range from 0-6. Higher scores indicate more frequent use of the respective strategies.
Coach Evaluations | Right after the intervention ended
  Goal attainment will be assessed by the coach using portions of the Goal Attainment Scaling (GAS) and therapy process scales (STEP-SV). Higher scores indicate higher goal achievement and better engagement.
Psychological distress | Baseline, right after the intervention ended, 3-month follow-up
  Somatization, depression, and anxiety syndromes will be assessed using the short version of the Brief Symptom Inventory (BSI-18). The total score on the BSI-18 is referred to as the Global Severity Index (GSI) and reflects the general psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive health information and cannot be sufficiently de-identified to ensure participant privacy. Data sharing is restricted by ethical approval and local data protection regulations.